CLINICAL TRIAL: NCT05668052
Title: A Cross-sectional Study of Covid-19 Pandemic in Zhejiang Province
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20221220,F1.0
Record Dates: First submitted 2022-12-28; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Cross-sectional Study; COVID-19 Pandemic
Keywords: Cross-sectional study; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — This survey was conducted in Zhejiang Provincial Hospital of Traditional Chinese Medicine from December 2022 to December 2023. The research objects were patients with COVID-19.

SUMMARY:
this study adopted a cross-sectional study, collected the medical history and symptoms of patients infected with Covid-19 through a questionnaire survey, and made statistical analysis, so as to provide better clinical guidance.

DETAILED DESCRIPTION:
Recently, there has been an outbreak of covid-19 in Zhejiang Province. In order to comprehensively understand the condition of patients with covid-19 in Zhejiang Province, this study adopted a cross-sectional study, collected the medical history and symptoms of patients infected with Covid-19 through a questionnaire survey, and made statistical analysis, so as to provide better clinical guidance.

ELIGIBILITY:
Inclusion Criteria:

* A positive nucleic acid test for Covid-19, or a positive antigen test for novel coronavirus, no age limit.

Exclusion Criteria:

* Unable to understand the contents of the questionnaire for various reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Covid-19
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-27 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
characters of patients with Covid-19 | baseline
  this study collected the medical history and symptoms of patients infected with Covid-19 through a questionnaire survey, and made statistical analysis